CLINICAL TRIAL: NCT00135928
Title: Bone Marrow Stimulation With G-CSF in Acute Myocardial Infarction,
Brief Title: Stem Cells in Myocardial Infarction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: STEMMI
Record Dates: First submitted 2005-08-25; First posted 2005-08-26 (Estimated); Last update posted 2011-08-08 (Estimated); Status verified 2005-02

CONDITIONS: Acute Myocardial Infarction
Keywords: ST-elevation myocardial infarction; granulocyte-colony stimulating factor angiogenesis; stem cells
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Filgrastim

INTERVENTIONS:
Drug: Granulocyte Colony Stimulating Factor G-CSF (Neupogen®)

SUMMARY:
The purpose of this trial is to investigate the effect of treatment with granulocyte-colony stimulating factor (G-CSF) bone marrow stimulation on circulating stem cells' ability to develop new blood vessels in the myocardium after an acute myocardial infarction.

DETAILED DESCRIPTION:
Intracoronary infusion of bone-marrow stem cells after a ST elevation myocardial infarction (STEMI) seems to improve cardiac function. An alternative strategy is increase of circulating stem cells by mobilisation from the bone marrow with Granulocyte-Colony Stimulating Factor (G-CSF).

Objective: To determine the short-term (30 days) safety of G-CSF therapy after a STEMI treated with acute percutaneous coronary intervention (PCI).

Methods: Patients with STEMI treated with PCI <12 hours after symptom onset were randomised (1:1) to G-CSF (10 μg/kg/d) or placebo for 6 days in a double-blind design. Other inclusion criteria: age 20-70 years, culprit lesion in a large coronary artery, and peak CKMB >100 microgram/L. Follow-up was done after 1, 5 and 6 months, with an angiogram at 5 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 20 and 70 years with STEMI were eligible if they had a successful PCI within 12 hours after onset of symptoms.
* The target lesion had to be located in the proximal section of the left anterior descending (LAD), left circumflex (LCX) or right coronary artery (RCA).
* Only patients with creatine kinase [CK]-MB >100 microgram/L or development of Q waves in the electrocardiogram were included.

Exclusion Criteria:

* Ventricular arrhythmia after PCI requiring treatment
* Pregnancy
* Unprotected left main stem lesion
* History of prior myocardial infarction
* Diagnosed or suspected cancer
* New York Heart Association (NYHA) class 3-4
* Known severe claustrophobia
* Significant stenosis in another coronary vessel than the acutely treated vessel, that might demand treatment with PCI or coronary artery bypass graft surgery (CABG) prior to the last follow-up exam.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78
Dates: Start 2003-05; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
The pre-specified primary endpoint is change in regional systolic wall thickening from day 1 to day 180 evaluated with cardiac magnetic resonance imaging (MRI)

SECONDARY OUTCOMES:
Change in ejection fraction, end-systolic and end-diastolic volumes, regional myocardial perfusion, and infarct size by MRI
Change in regional myocardial function by tissue Doppler echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Jens Kastrup, MD DMSc, Principal Investigator — 2014 Department of Cardiology, The Heart Centre, University Hospital Rigshospitalet, DK-2100 Copenhagen, Denmark.
Locations (1):
- 2014 Department of Cardiology, The Heart Centre, University Hospital Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Derived] Ripa RS, Jorgensen E, Kastrup J. Clinical outcome after stem cell mobilization with granulocyte-colony-stimulating factor after acute ST-elevation myocardial infarction: 5-year results of the STEMMI trial. Scand J Clin Lab Invest. 2013 Mar;73(2):125-9. doi: 10.3109/00365513.2012.750010. Epub 2013 Jan 3. PMID 23281844
- [Derived] Hedegaard A, Ripa RS, Johansen JS, Jorgensen E, Kastrup J. Plasma YKL-40 and recovery of left ventricular function after acute myocardial infarction. Scand J Clin Lab Invest. 2010 Apr;70(2):80-6. doi: 10.3109/00365510903518191. PMID 20102300
- [Derived] Overgaard M, Ripa RS, Wang Y, Jorgensen E, Kastrup J. Timing of granulocyte-colony stimulating factor treatment after acute myocardial infarction and recovery of left ventricular function: results from the STEMMI trial. Int J Cardiol. 2010 Apr 30;140(3):351-5. doi: 10.1016/j.ijcard.2008.11.120. Epub 2009 Jan 7. PMID 19131132